CLINICAL TRIAL: NCT03850665
Title: Comparison of Early Objective and Subjective Outcome in Patients After Hip Arthroplasty, Operated From Direct Anterior, Posterolateraland Anterolateral Approach: Prospective Randomized Clinical Trial
Brief Title: Comparison of Functional Outcome in Patients After Hip Arthroplasty Depending on Surgical Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Artur Stolarczyk, Head of the Department of Orthopaedics and Rehabilitation, Principal Investigator, Clinical Professor, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: THA/ Warsaw MU
Record Dates: First submitted 2018-09-15; First posted 2019-02-22 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Hip; Osteoarthritis
Keywords: total; hip; arthroplasty; surgical; approach
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Direct Anterior Approach (DAA) (Active Comparator): Direct Anterior Approach surgery to replace the hip.
  Interventions: Procedure: Direct Anterior Approach (DAA); Procedure: Anterolateral approach
- Anterolateral approach (Active Comparator): Anterolateral Approach surgery to replace the hip.
  Interventions: Procedure: Direct Anterior Approach (DAA); Procedure: Anterolateral approach
- Posterolateral approach (Active Comparator): Posterolateral Approach surgery to replace the hip.
  Interventions: Procedure: Direct Anterior Approach (DAA); Procedure: Anterolateral approach

INTERVENTIONS:
Procedure: Direct Anterior Approach (DAA) — Direct Anterior Approach surgery to replace the hip.
Procedure: Anterolateral approach — Anterolateral approach surgery to replace the hip.

SUMMARY:
The aim of the study will be to compare functional outcomes of the two surgical hip approaches in total hip arthroplasty: anterior, posterolateral and anterolateral. Surgical approach may have influence on patients functional outcome.

DETAILED DESCRIPTION:
Patients with primary hip osteoarthritis will be included in a randomized controlled trial and assigned to total hip arthroplasty using one the of hip approaches: anterior or anterolateral. Subjects will be assessed preoperative and 3 and 12 moths postoperative.

Biomechanical gait parameters will be collected using tree-dimensional motion analysis system "BTS SMART".

Evaluation of the function of the middle gluteal muscle with superficial EMG (sEMG) percutaneous surface electromyography. Fatigue assessment (mean frequency and amplitude) of the gluteus medius muscle during isometric muscle contraction.

Balance and coordination as well as fall risk will be assessed with use of dynamometric Biodex Balance platform. The study will determine the values of individual indicators: general stability index (OWS), anterior-posterior stability index (APW), the median lateral stability index (MLW) and the fall risk index (RU).

Subjective assessment will be conducted with use of Visual Analogue Scale, WOMAC Index, Oxford Hip Score, The Short Form-36 (SF-36) and Harris Hip Score

ELIGIBILITY:
Inclusion Criteria:

* patient's consent for anticipation in the study
* BMI less than 35
* ability to walk the distance of 10m and stand up from the chair
* arthroplasty in one hip

Exclusion Criteria:

* patient's lack of consent for anticipation in the study
* neurological diseases
* balance disorders
* reoperations in the area of endoprosthesis
* muscles diseases
* rheumatic diseases (rheumatoid arthritis, ankylosing spondylitis)
* dizziness, vasovagal syncope

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2020-09-27 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Change in biomechanical gait parameters | from baseline (can be measured anytime to a maximum of one month before surgery) to 3 and 12 months post-operatively
  Done by a biomechanics lab for patients to test their hip movements
Gluteus medius muscle fatigue | from baseline (can be measured anytime to a maximum of one month before surgery) to 3 and 12 months post-operatively
  Surface Electromyographic analysis performed for testing gluteus medius activity
Change from baseline in Hip disability and Osteoarthritis Outcome Score (HOOS) activities of daily living (ADL) | from baseline (can be measured anytime to a maximum of one month before surgery) to 3 and 12 months post-operatively
  This asks the patient how their hip functions during their daily life. It has 5 subscales measuring Pain, Symptoms, ADL, Sports/Recreation and Quality of Life (which is calculated using all the subscores). Each subscale is calculated using the mean score, with each score range being from 0 to 4. The subscore is normalized such that the lower the number the more extreme the problem is. To calculate Quality of Life, the mean of the other 4 subscores are taken to calculate the score.
  This asks the patient how their hip functions during their daily life. It has 5 subscales measuring Pain, Symptoms, ADL, Sports/Recreation and Quality of Life (which is calculated using all the subscores). Each subscale is calculated using the mean score, with each score range being from 0 to 4. The subscore is normalized such that the lower the number the more extreme the problem is. To calculate Quality of Life, the mean of the other 4 subscores are taken to calculate the score.
Change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | from baseline (can be measured anytime to a maximum of one month before surgery) to 3 and 12 months post-operatively
  This measures health status as it relates to the hip. There are 3 subscales, pain which score ranges from 0-20, stiffness range from 0-8, physical function ranging from 0-68. The total score is just added up from the subscales.
Change in Oxford scale | from baseline (can be measured anytime to a maximum of one month before surgery) to 3 and 12 months post-operatively
  The Oxford scale is a physiotherapist objective-rated scale to asses muscle strength against the resistance. It is graded from 0 (flicker of movement) to 5 (Through full range actively against strong resistance)
Change in SF-36 scale | from baseline (can be measured anytime to a maximum of one month before surgery) to 3 and 12 months post-operatively
  The SF-36 is a participant self-rated questionnaire that is a general measure of perceived health status comprising 36 questions, which yields an 8-scale health profile. The vitality sub-score assesses energy and fatigue, and ranges from 0 (worst) - 100 (best).
Change in Visual Analog Scale (VAS) scale | from baseline (can be measured anytime to a maximum of one month before surgery) to 3 and 12 months post-operatively
  To measure pain. This is a line with left most end representing no pain with the rightmost representing extreme pain. The participant puts a line where they feel that day and it is measured with a ruler to determine score out of 100. The line is 100mm long.
Change in biomechanical gait balance | from baseline (can be measured anytime to a maximum of one month before surgery) to 3 and 12 months post-operatively
  Done by a biomechanics lab for patients to test their gait balance
Change in biomechanical coordination | from baseline (can be measured anytime to a maximum of one month before surgery) to 3 and 12 months post-operatively
  Done by a biomechanics lab for patients to test their hip movements coordination

SECONDARY OUTCOMES:
Radiological analysis of implants positioning | from baseline (can be measured anytime to a maximum of one month before surgery) to 3 and 12 months post-operatively
  To measure angles associated with proper implants positioning

CONTACTS AND LOCATIONS:
Overall Officials: Artur Stolarczyk, Ph. D, Study Director — Orthopaedics and Rehabilitation Department, Medical University of Warsaw; Bartosz Maciąg, Principal Investigator — Orthopaedics and Rehabilitation Department, Medical University of Warsaw
Locations (2):
- Poland (2):
  - Department of Orthopedics and Rehabilitation, Medical University of Warsaw, Warsaw, Masovian Voivodeship
  - Orthopaedics and Rehabilitation Department, Medical University of Warsaw, Warsaw

REFERENCES:
- [Background] Mariconda M, Galasso O, Costa GG, Recano P, Cerbasi S. Quality of life and functionality after total hip arthroplasty: a long-term follow-up study. BMC Musculoskelet Disord. 2011 Oct 6;12:222. doi: 10.1186/1471-2474-12-222. PMID 21978244
- [Background] Sinha A, Twycross-Lewis R, Small C, Morrissey D, Maffulli N. Motion analysis as an outcome measure for hip arthroplasty. Surgeon. 2011 Oct;9(5):284-91. doi: 10.1016/j.surge.2011.02.002. Epub 2011 Mar 13. PMID 21843824
- [Background] Demos HA, Rorabeck CH, Bourne RB, MacDonald SJ, McCalden RW. Instability in primary total hip arthroplasty with the direct lateral approach. Clin Orthop Relat Res. 2001 Dec;(393):168-80. doi: 10.1097/00003086-200112000-00020. PMID 11764347
- [Background] Wylde V, Blom AW, Bolink S, Brunton L, Dieppe P, Gooberman-Hill R, Grimm B, Mann C, Lenguerrand E. Assessing function in patients undergoing joint replacement: a study protocol for a cohort study. BMC Musculoskelet Disord. 2012 Nov 13;13:220. doi: 10.1186/1471-2474-13-220. PMID 23148591
- [Background] Cheng TE, Wallis JA, Taylor NF, Holden CT, Marks P, Smith CL, Armstrong MS, Singh PJ. A Prospective Randomized Clinical Trial in Total Hip Arthroplasty-Comparing Early Results Between the Direct Anterior Approach and the Posterior Approach. J Arthroplasty. 2017 Mar;32(3):883-890. doi: 10.1016/j.arth.2016.08.027. Epub 2016 Aug 31. PMID 27687805
- [Background] Queen RM, Schaeffer JF, Butler RJ, Berasi CC, Kelley SS, Attarian DE, Bolognesi MP. Does surgical approach during total hip arthroplasty alter gait recovery during the first year following surgery? J Arthroplasty. 2013 Oct;28(9):1639-43. doi: 10.1016/j.arth.2013.02.008. Epub 2013 Mar 19. PMID 23518430
- [Background] Wesseling M, Meyer C, Corten K, Simon JP, Desloovere K, Jonkers I. Does surgical approach or prosthesis type affect hip joint loading one year after surgery? Gait Posture. 2016 Feb;44:74-82. doi: 10.1016/j.gaitpost.2015.11.009. Epub 2015 Nov 23. PMID 27004636
- [Background] Foucher KC, Wimmer MA, Moisio KC, Hildebrand M, Berli MC, Walker MR, Berger RA, Galante JO. Time course and extent of functional recovery during the first postoperative year after minimally invasive total hip arthroplasty with two different surgical approaches--a randomized controlled trial. J Biomech. 2011 Feb 3;44(3):372-8. doi: 10.1016/j.jbiomech.2010.10.026. Epub 2010 Nov 13. PMID 21075378
- [Background] Rosenlund S, Broeng L, Overgaard S, Jensen C, Holsgaard-Larsen A. The efficacy of modified direct lateral versus posterior approach on gait function and hip muscle strength after primary total hip arthroplasty at 12months follow-up. An explorative randomised controlled trial. Clin Biomech (Bristol). 2016 Nov;39:91-99. doi: 10.1016/j.clinbiomech.2016.09.011. Epub 2016 Sep 30. PMID 27721093
- [Background] Yue C, Kang P, Pei F. Comparison of Direct Anterior and Lateral Approaches in Total Hip Arthroplasty: A Systematic Review and Meta-Analysis (PRISMA). Medicine (Baltimore). 2015 Dec;94(50):e2126. doi: 10.1097/MD.0000000000002126. PMID 26683920
- [Background] Beaulieu ML, Lamontagne M, Beaule PE. Lower limb biomechanics during gait do not return to normal following total hip arthroplasty. Gait Posture. 2010 Jun;32(2):269-73. doi: 10.1016/j.gaitpost.2010.05.007. Epub 2010 Jun 11. PMID 20541940
- [Background] Bennett D, Humphreys L, O'Brien S, Kelly C, Orr JF, Beverland DE. Gait kinematics of age-stratified hip replacement patients--a large scale, long-term follow-up study. Gait Posture. 2008 Aug;28(2):194-200. doi: 10.1016/j.gaitpost.2007.11.010. Epub 2008 Feb 19. PMID 18242996
- [Background] Calo L, Rabini A, Picciotti PM, Laurino S, Passali GC, Ferrara PE, Maggi L, Piazzini DB, Specchia A, Frasca G, Ronconi G, Bertolini C, Scarano E. Postural control in patients with total hip replacement. Eur J Phys Rehabil Med. 2009 Sep;45(3):327-34. Epub 2009 Feb 11. PMID 19209135
- [Background] Soderman P, Malchau H, Herberts P. Outcome of total hip replacement: a comparison of different measurement methods. Clin Orthop Relat Res. 2001 Sep;(390):163-72. doi: 10.1097/00003086-200109000-00019. PMID 11550862
- [Background] McConnell S, Kolopack P, Davis AM. The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC): a review of its utility and measurement properties. Arthritis Rheum. 2001 Oct;45(5):453-61. doi: 10.1002/1529-0131(200110)45:53.0.co;2-w. No abstract available. PMID 11642645
- [Background] Kalairajah Y, Azurza K, Hulme C, Molloy S, Drabu KJ. Health outcome measures in the evaluation of total hip arthroplasties--a comparison between the Harris hip score and the Oxford hip score. J Arthroplasty. 2005 Dec;20(8):1037-41. doi: 10.1016/j.arth.2005.04.017. PMID 16376260
- [Background] Wylde V, Learmonth ID, Cavendish VJ. The Oxford hip score: the patient's perspective. Health Qual Life Outcomes. 2005 Oct 31;3:66. doi: 10.1186/1477-7525-3-66. PMID 16259627